CLINICAL TRIAL: NCT05098158
Title: Community-Engaged Options to Maximize and Facilitate Opioid Reduction Through Treatment
Brief Title: Community-Engaged Options to Facilitate Opioid Reduction
Acronym: COMFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Spokane Regional Health District (Unknown); University of Washington Institute for Translational Health Science (KL2) (Other); Rayce Rudeen Foundation (Unknown)
Responsible Party: Principal Investigator, Marian Wilson, Associate Professor, Washington State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18111
Record Dates: First submitted 2020-07-13; First posted 2021-10-28 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain
Keywords: chronic pain; opioid; complementary
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single group studied over 6 weeks time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm pain treatment (Experimental): Arm includes usual pain care plus the chosen two telehealth interventions x 6 weeks
  Interventions: Other: Non-pharmacological pain treatment

INTERVENTIONS:
Other: Non-pharmacological pain treatment — Participant selects from telehealth consultation on massage therapy, yoga therapy, chiropractic and physical therapies.

SUMMARY:
This study investigates how adults prescribed opioids for chronic noncancer pain respond to invitations to try non-opioid options of massage therapy, yoga therapy, chiropractic and physical therapies. Options will be available via telehealth consultation visits using a computer or smartphone with internet connection. The investigators will measure effects on pain, pain-related symptoms, and opioid use over time using a single-group design.

DETAILED DESCRIPTION:
Participants will be recruited from local primary care practices and asked to complete a baseline survey. They will then meet with a registered nurse via teleconference for a complete pain assessment. At the end of the session, participants will be asked to choose two of four available modalities for telehealth consultation. Participants will be scheduled for six telehealth sessions, once per week x six weeks with three consultations per each chosen therapy. Measurements of pain, mood, sleep, medicine use will be captured at baseline, three weeks and six weeks and examined for changes over time.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in treatment at the CHAS Perry St or partnering clinic;
* age greater than 18 years;
* ability to read, speak, and write English;
* diagnosed with a chronic, non-cancer-based painful medical condition;
* ability to provide informed consent.

Exclusion Criteria:

* pregnancy;
* diagnosis of a cancer-based painful medical condition;
* any other medical or psychiatric condition that the PI or Co-PI physician of record determine might compromise safe study participation (including but not limited to active psychosis, history of frequent psychiatric hospitalizations, severe anxiety with claustrophobia, aggression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Community Health Association of Spokane, Spokane, Washington
  - Washington State University College of Nursing, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Pain Treatment
Started | 16
Yoga Intervention | 11
Physical Therapy Intervention | 9
Massage Intevention | 8
Chiropractic Intervention | 4
Completed | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Pain Treatment
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
PROMIS Pain Intensity Scale [Mean (Standard Deviation); unit: units on a scale] — Full scale name is PROMIS (Patient-Reported Outcome Measurement Information System) Pain Intensity Scale version 3a that measures the construct pain intensity or severity in three items for how much it hurts on average, at its worst and at its least in the past 7 days. Scale ranges from minimum "no pain" =1 to maximum "very severe" =5 pain with a possible sum of 3-15. A total sum of the 3 items is converted into a T-score where 50 is equivalent to the U.S. general population average and + /- 10 points is equivalent to the standard deviation. Higher values are considered to be a worse outcome.
  units on a scale | 68.6 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Rating
Description: Full scale name is PROMIS (Patient-Reported Outcome Measurement Information System) Pain Intensity Scale version 3a that measures the construct pain intensity or severity in three items for how much it hurts on average, at its worst and at its least in the past 7 days. Scale ranges from minimum "no pain" =1 to maximum "very severe" =5 pain with a possible sum of 3-15. A total sum of the 3 items is converted into a T-score where 50 is equivalent to the U.S. general population average and + /- 10 points is equivalent to the standard deviation. Higher values are considered to be a worse outcome (range 40-70 after T-score conversion).
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Pain Treatment
Number analyzed (Participants) | 16
score on a scale
  Pre | 68.3 (6.3)
  Post: number analyzed (Participants) | 15
  Post | 64.4 (6.0)
Statistical Analysis 1: Comparison: Single Arm Pain Treatment; Paired t tests of pre and posttest data; Test type: Equivalence — Paired t tests had .05 set as level of significance to reject null hypothesis. Sample powered to generate effect size for future studies; p < 0.001, t-test, 2 sided — Actual p value results above; Not adjusted due to pilot study aim to generate effect size comparing pre and posttest data; Mean Difference (Final Values) = 3.9

2. Primary Outcome: PROMIS Pain Interference Rating
Description: Scale name is PROMIS (Patient-Reported Outcome Measurement Information System) Pain Interference Scale that measures the construct pain interference in 8 items for how much pain interferes with a variety of activities in the past 7 days. Scale ranges from minimum "not at all" =1 to maximum "very much" =5 pain with a possible sum of 8-40. A total sum of the 8 items is converted into a T-score where 50 is equivalent to the U.S. general population average and + /- 10 points is equivalent to the standard deviation. Higher values are considered to be a worse outcome.
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Pain Treatment
Number analyzed (Participants) | 16
units on a scale
  Pre | 69.9 (5.5)
  Post: number analyzed (Participants) | 15
  Post | 64.3 (8.3)
Statistical Analysis 1: Comparison: Single Arm Pain Treatment; Paired t tests of pre and posttest data; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.003, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.6

3. Secondary Outcome: Depressive Symptoms Using Patient Health Questionnaire (PHQ-8)
Description: Patient Health Questionnaire (PHQ-8) 8-item scale with score range 0-24 (higher score is worsened depressive symptoms)
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Pain Treatment
Number analyzed (Participants) | 16
score on a scale
  Pre | 10.7 (5.9)
  Post: number analyzed (Participants) | 15
  Post | 7.6 (5.0)
Statistical Analysis 1: Comparison: Single Arm Pain Treatment; Paired t tests of pre and posttest data; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.011, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.1

4. Secondary Outcome: PROMIS Self-efficacy for Managing Symptoms Short Form 4a
Description: Self-efficacy self-report (range 4-20 with higher score better symptom management self-efficacy). Scores converted into T scores with 50 as the average for US adults and + /- 10 points is equivalent to the standard deviation. Higher values are considered to be a better outcome (range 40-70 after T-score conversion).
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Pain Treatment
Number analyzed (Participants) | 16
units on a scale
  Pre | 39.4 (5.2)
  Post: number analyzed (Participants) | 15
  Post | 41.2 (5.3)
Statistical Analysis 1: Comparison: Single Arm Pain Treatment; Paired t tests of pre and posttest data; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.168, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.9

5. Secondary Outcome: PROMIS Self-efficacy for Managing Emotions Short Form 4a
Description: Self-efficacy self-report (range 4-20 ). Converted to T score where 50 equals the US adults average and + /- 10 points is equivalent to the standard deviation. Higher values are considered to be a better outcome for self-efficacy for managing emotions (range 40-70 after T-score conversion).
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Pain Treatment
Number analyzed (Participants) | 16
units on a scale
  Pre | 43.4 (6.3)
  Post: number analyzed (Participants) | 15
  Post | 44.4 (5.1)
Statistical Analysis 1: Comparison: Single Arm Pain Treatment; Paired t tests of pre and posttest data; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.456, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.1

6. Secondary Outcome: Anxiety Using Generalized Anxiety Disorder (GAD-7)
Description: 7-item scale with score range 0-21 (higher score is worsened anxiety)
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Single Arm: Participants with pre and post data for analysis
Arm/Group | Single Arm
Number analyzed (Participants) | 16
units on a scale
  Pre | 5.9 (4.7)
  Post: number analyzed (Participants) | 15
  Post | 5.2 (5.2)
Statistical Analysis 1: Comparison: Single Arm; Paired t tests of pre and posttest data; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.517, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = .8

7. Secondary Outcome: Interpersonal Needs Questionnaire
Description: 9-item scale asking how one feels about others score range 0-28 (lower score indicates more unmet interpersonal needs)
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 16
units on a scale
  Pre | 27.7 (14.4)
  Post: number analyzed (Participants) | 15
  Post | 24.5 (13.5)
Statistical Analysis 1: Comparison: Single Arm; Paired t tests of pre and posttest data; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.012, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.2

8. Secondary Outcome: Current Opioid Misuse Measure
Description: 17-item scale to ask about use of opioids (range 0-64 with higher scores indicating more misuse)
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 16
units on a scale
  Pre | 7.1 (4.9)
  Post: number analyzed (Participants) | 15
  Post | 6.8 (4.4)
Statistical Analysis 1: Comparison: Single Arm; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.811, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.3

9. Secondary Outcome: Spiritual Well-being Index
Description: 4-items to ask about spiritual well-being (range 4-20 with higher scores indicating more spiritual well-being)
Time Frame: 6 weeks
Population: Participants with pre and post data for analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 16
units on a scale
  Pre | 15 (4.1)
  Post: number analyzed (Participants) | 15
  Post | 15.1 (3.5)
Statistical Analysis 1: Comparison: Single Arm; Paired t tests of pre and posttest dat; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.941, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1

10. Other Pre Specified Outcome: Percentage of Attendance in Scheduled Telehealth Sessions
Description: Percentage of scheduled telehealth sessions attended by participants (calculated as total number attended/total number scheduled)
Time Frame: 6 weeks
Population: All participants
Measure: Number; unit: percentage of sessions attended
Units Other Than Participants: telehealth sessions
Groups:
- Single Arm: All participants
Arm/Group | Single Arm
Number analyzed (Participants) | 16
Number analyzed (telehealth sessions) | 96
percentage of sessions attended | 95.8
Statistical Analysis 1: Comparison: Single Arm; Test type: Other — Descriptive statistics to report the percentage of offered telehealth sessions that were attended [#attended/#offered = % attended]; percentage = 95.8

11. Other Pre Specified Outcome: IBM Computer Usability and Satisfaction Questionnaires
Description: The IBM Computer Usability and Satisfaction Questionnaires was adapted to measure tele-visit program usability and satisfaction with a 4-item survey to gauge participant satisfaction with the intervention using 1-7 Likert scale. A total mean satisfaction rating was generated from the combined mean 4 satisfaction items (possible mean range 1-7 where higher score means higher satisfaction) on a Likert-style scale: The Likert-style scale for each item was: 1: Strongly disagree- 7: Strongly agree where higher numbers indicate greater satisfaction.
Time Frame: 6 weeks
Population: Participants with satisfaction data completed - 1 did not participate
Measure: Mean (Standard Deviation); unit: mean of summed scores on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 15
mean of summed scores on a scale | 6.59 (0.62)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Severity of event was rated as (select one): Grade 1 - Mild; Grade 2 - Moderate; Grade 3 - Severe Participants were evaluated by RN as to whether there was a reasonable possibility that the experimental COMFORT intervention caused the event.
Arm/Group | Single Arm Pain Treatment
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Pain Treatment (N=16)
Mild (Ear and labyrinth disorders) | 1 (1) — Vertigo reported by participant; does not believe it was related to the study intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05098158/Prot_SAP_ICF_000.pdf